CLINICAL TRIAL: NCT05658042
Title: Therapeutic Drug Monitoring Combined With Quantitative Pharmacology for Dose Optimization of Rivaroxaban in Combination With Rifampicin in Patients With Periprosthetic Joint Infection
Brief Title: Dose Optimization of Rivaroxaban Combined With Rifampicin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-LCYJ-PY-41
Record Dates: First submitted 2022-11-27; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-03

CONDITIONS: Infections
Keywords: periprosthetic infection; rivaroxaban
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- rivaroxaban 10mg qd: nonintervention
- rivaroxaban 10mg qd+rifampicin: nonintervention
- rivaroxaban 20mg qd+rifampicin: nonintervention
- rivaroxaban 15mg bid+rifampicin: nonintervention

SUMMARY:
The goal of this observational study is to learn about exposure levels of rivaroxaban at different doses in patients with prosthetic joint infection combined with the use of rifampicin. Participants will be collected blood samples to determine rivaroxaban plasma concentration. The main question it aims to answer is to predict the dose adjustment of rivaroxaban combined with the use of rifampin.

DETAILED DESCRIPTION:
This study is a prospective observational study and does not interfere with the normal clinical diagnosis and treatment process. In the case of patients with periprosthetic infection with or without rifampicin, the blood concentration of rivaroxaban was monitored, and the data were further predicted and analyzed by statistical tests and physiological pharmacokinetic models, and suggestions were made for dose optimization.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged>18 years
* The diagnosis was periprosthetic infection after joint replacement
* Orthopedic operations such as revision of artificial joints, removal of prostheses, debridement, etc. for the treatment of periprosthetic infection
* Rivaroxaban was used to prevent deep vein thrombosis after operation.

Exclusion Criteria:

* Patients allergic to any excipient in rivaroxaban, rifampicin or tablets
* Patients with clinically significant active bleeding
* Patients with significant risk of bleeding
* Patients with liver disease with coagulation abnormalities and clinical-related bleeding risk, including patients with cirrhosis who reached Child Pugh C grade
* Pregnant women and breastfeeding women
* Patients taking combined drugs affecting rivaroxaban metabolism
* Patients who were unable or unwilling to cooperate with the study (Such as mental or memory disorders)
* Patients discontinued without meeting study target days
* Patients with severe renal insufficiency (creatinine clearance rate < 30ml / min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
plasma concentration of rivaroxaban | 2-4 hours and 12-16 hours after 2-5 days of continuous dosing for rivaroxaban
  HPLC-MS/MS method

SECONDARY OUTCOMES:
incidence of adverse reactions | From admission to discharge, up to 3 week
  Bleeding and anemia
effect indicator | From admission to discharge, up to 3 week
  Activated Partial Thromboplastin Time and Prothrombin time

CONTACTS AND LOCATIONS:
Overall Officials: Ruijuan Xu, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falck-Ytter Y, Francis CW, Johanson NA, Curley C, Dahl OE, Schulman S, Ortel TL, Pauker SG, Colwell CW Jr. Prevention of VTE in orthopedic surgery patients: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e278S-e325S. doi: 10.1378/chest.11-2404. PMID 22315265
- [Background] Gnoth MJ, Buetehorn U, Muenster U, Schwarz T, Sandmann S. In vitro and in vivo P-glycoprotein transport characteristics of rivaroxaban. J Pharmacol Exp Ther. 2011 Jul;338(1):372-80. doi: 10.1124/jpet.111.180240. Epub 2011 Apr 22. PMID 21515813
- [Background] Lang D, Freudenberger C, Weinz C. In vitro metabolism of rivaroxaban, an oral, direct factor Xa inhibitor, in liver microsomes and hepatocytes of rats, dogs, and humans. Drug Metab Dispos. 2009 May;37(5):1046-55. doi: 10.1124/dmd.108.025551. Epub 2009 Feb 5. PMID 19196846
- [Background] Weinz C, Schwarz T, Kubitza D, Mueck W, Lang D. Metabolism and excretion of rivaroxaban, an oral, direct factor Xa inhibitor, in rats, dogs, and humans. Drug Metab Dispos. 2009 May;37(5):1056-64. doi: 10.1124/dmd.108.025569. Epub 2009 Feb 5. PMID 19196845
- [Background] Osmon DR, Berbari EF, Berendt AR, Lew D, Zimmerli W, Steckelberg JM, Rao N, Hanssen A, Wilson WR; Infectious Diseases Society of America. Diagnosis and management of prosthetic joint infection: clinical practice guidelines by the Infectious Diseases Society of America. Clin Infect Dis. 2013 Jan;56(1):e1-e25. doi: 10.1093/cid/cis803. Epub 2012 Dec 6. PMID 23223583
- [Background] Vakkalagadda B, Frost C, Byon W, Boyd RA, Wang J, Zhang D, Yu Z, Dias C, Shenker A, LaCreta F. Effect of Rifampin on the Pharmacokinetics of Apixaban, an Oral Direct Inhibitor of Factor Xa. Am J Cardiovasc Drugs. 2016 Apr;16(2):119-27. doi: 10.1007/s40256-015-0157-9. PMID 26749408
- [Background] Altena R, van Roon E, Folkeringa R, de Wit H, Hoogendoorn M. Clinical challenges related to novel oral anticoagulants: drug-drug interactions and monitoring. Haematologica. 2014 Feb;99(2):e26-7. doi: 10.3324/haematol.2013.097287. No abstract available. PMID 24497568
- [Background] Becerra AF, Amuchastegui T, Tabares AH. Decreased Rivaroxaban Levels in a Patient with Cerebral Vein Thrombosis Receiving Phenytoin. Case Rep Hematol. 2017;2017:4760612. doi: 10.1155/2017/4760612. Epub 2017 Aug 10. PMID 28875044
- [Background] Mueck W, Borris LC, Dahl OE, Haas S, Huisman MV, Kakkar AK, Kalebo P, Muelhofer E, Misselwitz F, Eriksson BI. Population pharmacokinetics and pharmacodynamics of once- and twice-daily rivaroxaban for the prevention of venous thromboembolism in patients undergoing total hip replacement. Thromb Haemost. 2008 Sep;100(3):453-61. PMID 18766262
- [Background] Wyse DG. Targeted Therapeutic Drug Monitoring for Direct Oral Anticoagulants: What Is Its Potential Place and Can It Limit Black Swan Events? Can J Cardiol. 2018 Nov;34(11):1393-1395. doi: 10.1016/j.cjca.2018.08.006. Epub 2018 Aug 9. No abstract available. PMID 30404744
- [Background] Bernier M, Lancrerot SL, Parassol N, Lavrut T, Viotti J, Rocher F, Drici MD. Therapeutic Drug Monitoring of Direct Oral Anticoagulants May Increase Their Benefit-Risk Ratio. J Cardiovasc Pharmacol. 2020 Oct;76(4):472-477. doi: 10.1097/FJC.0000000000000870. PMID 33030858
- [Background] Min JS, Bae SK. Prediction of drug-drug interaction potential using physiologically based pharmacokinetic modeling. Arch Pharm Res. 2017 Dec;40(12):1356-1379. doi: 10.1007/s12272-017-0976-0. Epub 2017 Oct 27. PMID 29079968